CLINICAL TRIAL: NCT05737927
Title: Pharmacodynamics and Pharmacokinetics of Different Coated and Uncoated Formulations of Glucose Beads After Single and Multiple Dose Administration Under Fasting Conditions in Obese Healthy Subjects
Brief Title: Pharmacodynamics and Pharmacokinetics of Different Glucose Bead Formulations in Obese Healthy Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Aphaia Pharma US LLC (Industry)
Collaborators: NovaClin Medical Research Center S.R.L (Unknown); ACC GmbH Analytical Clinical Concepts (Unknown); SC Bioclinica SA (Unknown); Galephar Pharmaceutical Research (PR), Inc. (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 008B20
Record Dates: First submitted 2023-01-19; First posted 2023-02-21 (Actual); Last update posted 2025-09-18 (Actual); Status verified 2025-09

CONDITIONS: Obese
MeSH Terms: conditions — Obesity | interventions — Glucose

STUDY DESIGN:
Intervention Model Description: Part 1: randomised, open label, five-treatment, five-period, five-sequence, crossover, at one study site
  Part 2: open label, one-treatment, one-period, at one study site
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (6):
- SINGLE DOSE- TEST PRODUCT 1 (T1) (Active Comparator): Oral coated beads 8 g glucose (content glucose/bead 47% w/w)
  Interventions: Drug: Glucose 8 g coated beads (47% w/w)
- SINGLE DOSE- TEST PRODUCT 2 (T2) (Active Comparator): Oral coated beads 12 g glucose (content glucose/bead 47% w/w)
  Interventions: Drug: Glucose 12 g coated beads (47% w/w)
- SINGLE DOSE- TEST PRODUCT 3 (T3) (Active Comparator): Oral coated beads 16 g glucose (content glucose/bead 47% w/w)
  Interventions: Drug: Glucose 16 g coated beads (47% w/w)
- SINGLE DOSE- TEST PRODUCT 4 (T4) (Active Comparator): Oral uncoated beads 12 g glucose
  Interventions: Drug: Glucose 12 g uncoated beads
- SINGLE DOSE- TEST PRODUCT 5 (T5) (Active Comparator): Oral coated beads 12 g glucose (content glucose/bead 60% w/w)
  Interventions: Drug: Glucose 12 g coated beads (60% w/w)
- MULTIPLE DOSE- TEST PRODUCT 2 (T2) (Active Comparator): Oral coated beads 12 g glucose (content glucose/bead 47% w/w)
  Interventions: Drug: Glucose 12 g coated beads (47% w/w)

INTERVENTIONS:
Drug: Glucose 8 g coated beads (47% w/w) — After an overnight fasting of about 10 hours, the subjects were administered 8 g glucose of the coated Glucose beads formulation starting at 8:00 (time 0; administration time was staggered beginning at 8:00 for the first group of subjects) in sitting position.
  Other Names: APHD-008
  Arms: SINGLE DOSE- TEST PRODUCT 1 (T1)
Drug: Glucose 12 g coated beads (47% w/w) — After an overnight fasting of about 10 hours, the subjects were administered 12 g glucose of the coated Glucose beads formulation starting at 8:00 (time 0; administration time was staggered beginning at 8:00 for the first group of subjects) in sitting position.
  Other Names: APHD-012
  Arms: SINGLE DOSE- TEST PRODUCT 2 (T2)
Drug: Glucose 16 g coated beads (47% w/w) — After an overnight fasting of about 10 hours, the subjects were administered 16 g glucose of the coated Glucose beads formulation starting at 8:00 (time 0; administration time was staggered beginning at 8:00 for the first group of subjects) in sitting position.
  Other Names: APHD-016
  Arms: SINGLE DOSE- TEST PRODUCT 3 (T3)
Drug: Glucose 12 g uncoated beads — After an overnight fasting of about 10 hours, the subjects were administered the uncoated Glucose beads formulation containing 12 g glucose starting at 8:00 (time 0; administration time was staggered beginning at 8:00 for the first group of subjects) in sitting position.
  Other Names: APHD-012P
  Arms: SINGLE DOSE- TEST PRODUCT 4 (T4)
Drug: Glucose 12 g coated beads (60% w/w) — After an overnight fasting of about 10 hours, the subjects were administered the coated Glucose beads formulation (60 % w/w glucose/bead; 12 g glucose) starting at 8:00 (time 0; administration time was staggered beginning at 8:00 for the first group of subjects) in sitting position.
  Other Names: APHD-012-60
  Arms: SINGLE DOSE- TEST PRODUCT 5 (T5)
Drug: Glucose 12 g coated beads (47% w/w) — After an overnight fasting of at least 10 hours, the subjects were administered the new developed Glucose beads formulation containing 12 g glucose starting at 8:00 (time 0; administration time was staggered beginning at 8:00 for the first group of subjects) in sitting position. Treatment duration: Day 1 - Day 4
  Other Names: APHD-012
  Arms: MULTIPLE DOSE- TEST PRODUCT 2 (T2)

SUMMARY:
The goal of this clinical study was to assess pharmacodynamics (PD) and pharmacokinetics (PK) of different Glucose beads formulations in obese healthy subjects under fasting condition. The study was designed in 2 parts.

Part 1 (single-dose) of the study was randomized, open label, five-treatment, five-period, five-sequence, crossover and single-centric. Treatment arms were three dosages of a coated Glucose beads formulation (47% w/w glucose/bead; 8 g [T1], 12 g [T2] and 16 g glucose [T3]), one uncoated Glucose beads formulation (47% w/w glucose/bead; 12 g glucose [T4]) and one coated Glucose beads formulation (60% w/w glucose/bead;12 g glucose [T5]).

Part 2 (multiple-dose) of the study was open label, one-treatment, one-period and single-centric. Treatment arm was coated Glucose beads formulation (12 g glucose [T2]).

DETAILED DESCRIPTION:
Twenty healthy obese subjects were planned for this study. Eligible subjects fulfilling the inclusion/ exclusion criteria and who had willing to give their informed consent were enrolled for screening examination and, if found eligible, enrolled in the study.

Before each hospitalization, on day -1, subjects with Real-Time Reverse Transcription-Polymerase Chain Reaction (rRT-PCR) tested negative for the new severe acute respiratory syndrome coronavirus 2 (SARS-CoV-2) coronavirus were hospitalized. At the hospitalization examination physical examinations (weight), vital signs, pregnancy test for female subjects, alcohol breath test, as well as a check of adverse events, inclusion and exclusion criteria and restrictions were performed. Subjects were admitted to the clinical site at least 13 hours prior to the administration of investigational product in each treatment period.

During each treatment period the hospitalization period in the clinical unit was 13 hours before and up to 11 hours after investigational product administration. Part 1: Single dose After an overnight fasting of at least 10 hours the subjects was administered either 8 g glucose (T1), 12 g glucose (T2), 16 g glucose (T3) of the coated Glucose beads formulation (47%), the uncoated Glucose beads formulation (T4) containing 12 g glucose (47%) or the coated Glucose beads formulation (60% w/w glucose/bead; 12 g glucose [T5]) starting at 8:00 (time 0; administration time was staggered beginning at 8:00 for the first group of subjects) in sitting position.

17 blood samples was drawn for determination of glucagon-like polypeptide 1 (GLP-1) levels at the prescribed times pre-dose (-1.0 h, -0.5 and 0.0 h [within 5 minutes]) and 0.5, 1.0, 1.5. 2.0, 2.5, 3.0, 3.5, 4.0, 4.5, 5.0. 5.5, 6.0, 8.0 and 10.0 hours after investigational product administration.

A fraction of one pre-dose sample (-1.0 h) before investigational product administration in treatment period I was also used to determine circulating concentration of microRNA (miRNA) 1983.

One additional blood sample was drawn pre-dose (-1.0 h) before investigational product administration in treatment period I for determination of adiponectin level.

Fractions of the blood samples was also used to determine circulating concentrations of 13 diabetes and obesity related hormones and inflammatory proteins (amylin c-peptide, ghrelin, gastric inhibitory polypeptide [GIP], GLP-1, glucagon, interleukin-6 [IL-6], insulin, leptin, monocyte chemoattractant protein-1 [MCP-1], pancreatic polypeptide [PP], peptide tyrosine tyrosine [PYY], tumor necrosis factor alpha [TNFa]) with formulation T3 (16 g glucose).

Part 2: Multiple dose After an overnight fasting of at least 10 hours, the subjects were administered the new developed Glucose beads formulation containing 12 g glucose starting at 8:00 (time 0: administration time was be staggered beginning at 8.00 for the first group of subjects) in sitting position for the 3 days.

Standard meals were provided 0.5 h (morning meal), 4.5 h (mid-day meal) and 10 h (evening meal) after investigational product administration.

Blood samples were drawn for determination of GLP-1 levels before (-1.0 h, -0.5 h and 0 h [within 5 minutes]) each investigational product administration (total 9 samples) on each day.

Venous blood glucose measurement was performed before each investigational product administration (total 3 samples).

On Day 4, after an overnight fasting of at least 10 hours the subjects were administered the Glucose beads formulation containing 12 g glucose starting at 8:00 (time 0; administration time was staggered beginning at 8:00 for the first group of subjects) in sitting position.

17 blood samples were drawn for determination of GLP-1 levels at the prescribed times pre-dose (-1.0 h, -0.5 h and 0 h [within 5 minutes]) and 0.5, 1.0, 1.5, 2.0, 2.5, 3.0, 3.5, 4.0, 4.5, 5.0, 5.5, 6.0, 8.0 and 10.0 hours after investigational product administration.

A fraction of one blood sample (10.0 h) was also used to determine circulating concentrations of miRNA1983.

One additional blood sample was drawn (10.0 h) for determination of adiponectin level.

Fractions of the blood samples was also used to determine circulating concentrations of 13 diabetes and obesity related hormones and inflammatory proteins (amylin c-peptide, ghrelin, GIP, GLP-1, glucagon, IL-6, insulin, leptin, MCP-1, PP, PYY, TNFa).

Follow-up Within 7 days after last blood sampling in the last treatment period, 12-lead ECG, clinical routine laboratory parameters, vital signs (blood pressure, heart rate, body temperature) and physical examination were repeated. Furthermore questioning for subjective well-being and questioning of adverse events was performed.

Wash-out periods Wash-out periods of at least 3 days separated the five treatment periods. A wash-out period of at least 3 days separated part 1 (single dose) and part 2 (multiple dose) of the study.

ELIGIBILITY:
Inclusion Criteria:

* Healthy obese, Caucasian, male and female subjects 18 - 55 years of age
* Body mass index within the range of > 30.0 kg/m2
* Waist circumference: men > 102 cm
* women > 88 cm
* Female subjects of childbearing potential agree to undergo pregnancy tests and to use an appropriate method of contraception (i.e. oral contraceptive steroids, intrauterine device, barrier method)
* Findings within the range of clinical acceptability in medical history (or the clinical investigator considers the deviation to be irrelevant for the purpose of the study)
* Findings within the range of clinical acceptability in physical examination (or the clinical investigator considers the deviation to be irrelevant for the purpose of the study)
* Laboratory values within the normal range (or the clinical investigator considers the deviation to be irrelevant for the purpose of the study)
* Normal ECG or abnormalities which the clinical investigator does not consider a disqualification for participation in the study
* Normal vital signs (normal blood pressure and heart rate measured under stabilised conditions at screening visit after at least 5 minutes of rest in sitting position) or abnormalities which the clinical investigator does not consider a disqualification for participation in the study
* Normal GI function, or abnormalities which the clinical investigator does not consider a disqualification for participation in the study
* Willingness to undergo screening and follow-up examinations (i.e. physical examinations and laboratory investigations before and after the treatment periods)
* Ability to comprehend subject information and willingness to sign the informed consent

Exclusion Criteria:

* Gastrointestinal, hepatic and renal diseases and/or pathological findings, which might interfere with pharmacokinetics and pharmacodynamics of the investigational product
* Established diagnosis of type-1 or type-2 diabetes mellitus
* Treatment with insulin, insulin secretagogues (sulfonylurea derivatives, glinides, GLP-1 agonists (exenatide, lixisenatide, glutides), or thiazolidinediones (glitazones)
* Unexplained rise in blood glucose
* Treatment for constipation (including but not limited to lactulose or any other form of stool softeners, laxatives) or diarrhea (including but not limited to pectins, loperamide etc.) or any other medication known to interfere with gastrointestinal transit time, such as e.g. metoclopramide, opioids, or gastric potential of hydrogen (pH) (including but not limited to antacids, H2-receptor antagonists, prazoles)
* History of hypersensitivity to the investigational product or any related drugs or to any of the excipients
* History or presence of any clinically significant cardiovascular, pulmonary, hepatobiliary, renal, hematological, gastrointestinal, endocrinologic, immunologic, dermatologic, neurological, psychiatric, metabolic, musculoskeletal, or malignant disease, which the clinical investigator does not consider a disqualification for participation in the study
* Known heart failure (Grade I to IV of New York Heart Association classification)
* Significant renal disease, including nephritic syndrome, chronic renal failure (defined as creatinine clearance < 60 mL/min and serum creatinine >180 μmol/L)
* Unexplained serum creatine phosphokinase (CPK) > 3-times the upper limit of normal (ULN).
* Subjects with a reason for CPK elevation may have the measurement repeated prior to randomization; a CPK retest > 3-times ULN leads to exclusion.
* Clinically significant abnormal laboratory values
* Clinically significant ECG findings
* Clinically significant vital signs
* Clinically significant illness or surgery within 4 weeks prior to dosing
* Less than 14 days after last acute disease
* Volunteers liable to orthostatic dysregulation, fainting, or blackouts
* History of, or current compulsive alcohol abuse (more than a total of 10 drinks weekly whereby one drink corresponds to 500 ml beer, 200 ml wine or 50 g spirits); or regular exposure to other substances of abuse
* Donation or loss of blood equal to or exceeding 500 ml during 90 days before the first administration of investigational product
* Positive testing for human immunodeficiency virus (HIV), hepatitis B surface antigen (HBsAg) and hepatitis C-virus (HCV)
* Participation in another study with an experimental drug within at least 3 months (or within five elimination half-lives of the previous experimental drug, whichever is longer) before the first administration of investigational product
* Any use of drug, prescribed or over the counter (OTC) (inclusive herbal remedies), within 2 weeks (or within six elimination half-lives of this medication, whichever is longer) prior to the first administration of investigational product except if this will not affect the outcome of the study in the opinion of the clinical investigator
* Pregnant women (positive pregnancy test)
* Lactating women
* Failure to provide informed consent
* Unwillingness or inability to comply with the study protocol or study-related procedures (e.g. difficulty to stay fasting, consume the standard meals, or swallow the beads formulations; difficult venous access)
* Positive result of rRT-PCR test to detect infection with the new SARS-CoV-2 coronavirus

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20 (Actual)
Dates: Start 2020-09-16 (Actual); Primary Completion 2020-11-09 (Actual); Study Completion 2020-11-09 (Actual)

PRIMARY OUTCOMES:
GLP-1 | Pre-dose (-1.0 hour, -0.5 hour and 0 hour [within 5 minutes]) and 0.5, 1.0, 1.5, 2.0, 2.5, 3.0, 3.5, 4.0, 4.5, 5.0, 5.5, 6.0, 8.0 and 10.0 hours after investigational product administration.
  Part 1: Area under the plasma concentration-time curve from the first time point zero to the last measured concentration (AUC[0-t])
GLP-1 | Pre-dose (-1.0 hour, -0.5 hour and 0 hour [within 5 minutes]) and 0.5, 1.0, 1.5, 2.0, 2.5, 3.0, 3.5, 4.0, 4.5, 5.0, 5.5, 6.0, 8.0 and 10.0 hours after investigational product administration.
  Part 1: Area under the plasma concentration-time curve from the time point 1.5 hours to 8 hours (AUC[1.5 hours-8 hours])
GLP-1 | Pre-dose (-1.0 hour, -0.5 hour and 0 hour [within 5 minutes]) and 0.5, 1.0, 1.5, 2.0, 2.5, 3.0, 3.5, 4.0, 4.5, 5.0, 5.5, 6.0, 8.0 and 10.0 hours after investigational product administration.
  Part 1: Adjusted area under the plasma concentration-time curve from the time point 1.5 hours to 8 hours (AUCadj.[1.5 hours-8 hours])
GLP-1 | Pre-dose (-1.0 hour, -0.5 hour and 0 hour [within 5 minutes]) and 0.5, 1.0, 1.5, 2.0, 2.5, 3.0, 3.5, 4.0, 4.5, 5.0, 5.5, 6.0, 8.0 and 10.0 hours after investigational product administration.
  Part 1: Maximum plasma concentration (Cmax[0-t])
GLP-1 | Pre-dose (-1.0 hour, -0.5 hour and 0 hour [within 5 minutes]) and 0.5, 1.0, 1.5, 2.0, 2.5, 3.0, 3.5, 4.0, 4.5, 5.0, 5.5, 6.0, 8.0 and 10.0 hours after investigational product administration.
  Part 1: Maximum plasma concentration between the time point 1.5 hours to 8 hours (Cmax[1.5 hours-8 hours])
GLP-1 | Pre-dose (-1.0 hour, -0.5 hour and 0 hour [within 5 minutes]) and 0.5, 1.0, 1.5, 2.0, 2.5, 3.0, 3.5, 4.0, 4.5, 5.0, 5.5, 6.0, 8.0 and 10.0 hours after investigational product administration.
  Part 1: Adjusted maximum plasma concentration between the time point 1.5 hours to 8 hours (Cmax,adj.[1.5 hours-8 hours])
GLP-1 | Pre-dose (-1.0 hour, -0.5 hour and 0 hour [within 5 minutes]) and 0.5, 1.0, 1.5, 2.0, 2.5, 3.0, 3.5, 4.0, 4.5, 5.0, 5.5, 6.0, 8.0 and 10.0 hours after investigational product administration.
  Part 1: Time of maximum plasma concentration (tmax[0-t])
GLP-1 | Pre-dose (-1.0 hour, -0.5 hour and 0 hour [within 5 minutes]) and 0.5, 1.0, 1.5, 2.0, 2.5, 3.0, 3.5, 4.0, 4.5, 5.0, 5.5, 6.0, 8.0 and 10.0 hours after investigational product administration.
  Part 1: Time of maximum plasma concentration between the time point 1.5 hours to 8 hours (tmax[1.5 hours-8 hours])
GLP-1 | Day 1-3:- pre-dose (-1.0 hour, -0.5 hour and 0 hour). Day 4:- Pre-dose (-1.0 hour, -0.5 hour and 0 hour [within 5 minutes]) and 0.5, 1.0, 1.5, 2.0, 2.5, 3.0, 3.5, 4.0, 4.5, 5.0, 5.5, 6.0, 8.0 and 10.0 hours after investigational product administration.
  Part 2: Area under the plasma concentration-time curve during a dosage interval at steady state (AUC[0-τ])
GLP-1 | Day 1-3:- pre-dose (-1.0 hour, -0.5 hour and 0 hour). Day 4:- Pre-dose (-1.0 hour, -0.5 hour and 0 hour [within 5 minutes]) and 0.5, 1.0, 1.5, 2.0, 2.5, 3.0, 3.5, 4.0, 4.5, 5.0, 5.5, 6.0, 8.0 and 10.0 hours after investigational product administration.
  Part 2: Maximum plasma concentration at steady state (Cmax,ss)
GLP-1 | Day 1-3:- pre-dose (-1.0 hour, -0.5 hour and 0 hour). Day 4:- Pre-dose (-1.0 hour, -0.5 hour and 0 hour [within 5 minutes]) and 0.5, 1.0, 1.5, 2.0, 2.5, 3.0, 3.5, 4.0, 4.5, 5.0, 5.5, 6.0, 8.0 and 10.0 hours after investigational product administration.
  Part 2: Concentration at the end of the dosing interval at steady state (Cτ,ss)

SECONDARY OUTCOMES:
Glucose levels | Pre-dose (-1.0 hour, 0 hour [within 5 minutes]) and 0.5, 1.0, 2.0, 3.0, 4.0, 5.0, 6.0, 8.0 and 10.0 hours after investigational product administration.
  Part 1: AUC(0-t)
Glucose levels | Pre-dose (-1.0 hour, 0 hour [within 5 minutes]) and 0.5, 1.0, 2.0, 3.0, 4.0, 5.0, 6.0, 8.0 and 10.0 hours after investigational product administration.
  Part 1: Cmax
Glucose levels | Day 1- Day 3:- Pre-dose (3 samples). Day 4:- Pre-dose (-1.0 hour, 0 hour [within 5 minutes]) and 0.5, 1.0, 2.0, 3.0, 4.0, 5.0, 6.0, 8.0 and 10.0 hours after investigational product administration.
  Part 2: Minimum blood concentration at steady state (Cmin,ss)
Glucose levels | Day 1- Day 3:- Pre-dose (3 samples). Day 4:- Pre-dose (-1.0 hour, 0 hour [within 5 minutes]) and 0.5, 1.0, 2.0, 3.0, 4.0, 5.0, 6.0, 8.0 and 10.0 hours after investigational product administration.
  Part 2: Time of maximum blood concentration at steady state (tmax,ss)
Visual analogue scale appetite | Pre-dose (0 hour) and 2, 3, 4, 5, 6, 8 and 10 hours after investigational product administration.
  Visual analogue scale for appetite ranges from 0 - 10. 0 represents very weak appetite while 10 represent very strong appetite.
Visual analogue scale stomach rumbles | Pre-dose (0 hour) and 2, 3, 4, 5, 6, 8 and 10 hours after investigational product administration.
  Visual analogue scale for stomach rumbles ranges from 0 - 10. 0 represents not hungry at all while 10 represent as hungry as I have ever felt.

CONTACTS AND LOCATIONS:
Overall Officials: Carmen Vizman, Principal Investigator — NovaClin Medical Research Center S.R.L
Locations (1):
- NovaClin Medical Research Center S.R.L, Timișoara, Romania, Romania

IPD SHARING:
Plan to Share IPD: No